CLINICAL TRIAL: NCT05941351
Title: fixAtion of skiN Flaps After Mastectomy Using ruNning or Interrupted suturEs for Combatting Seroma
Acronym: ANNIE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: METCZ20230049
Record Dates: First submitted 2023-07-03; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-06

CONDITIONS: Seroma
MeSH Terms: conditions — Seroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Running (Other): Group 1: Flap fixation after mastectomy with running sutures.
  Interventions: Procedure: flap fixation
- Individual (Other): Group 2: Flap fixation after mastectomy with interrupted sutures.
  Interventions: Procedure: flap fixation

INTERVENTIONS:
Procedure: flap fixation — flap fixation using running or interrupted sutures

SUMMARY:
Rationale: Flap fixation significantly reduces the incidence of seroma formation after mastectomy. Therefore, research should focus on finding the most optimal way to secure the skin flaps to the pectoral muscle. Previous studies have compared running sutures, interrupted sutures and tissue glue application to conventional wound closure. A recent systematic review with network meta-analysis indicated running sutures as the most optimal technique, however direct comparisons and high quality articles were lacking.

Objective: This prospective trial aims to directly compare running sutures with interrupted sutures in order to prevent complications in patients undergoing a mastectomy.

Study design: This trial will combine a retrospective cohort from the previous SARA-trial in Zuyderland MC with a randomised prospective trial. This study design was chosen to acquire a sample size with sufficient power and the ability to conduct this study in an acceptable time frame.

Study population: A retrospective cohort of patients participating in the SARA trial (RCT) and a prospective cohort of patients undergoing a mastectomy for breast cancer.

Intervention: Group 1: Flap fixation after mastectomy with running sutures. Group 2: Flap fixation after mastectomy with interrupted sutures.

Main study parameters/endpoints: The primary endpoint is the incidence of complications requiring interventions in both groups, including clinically significant seroma, infections and bleeding complications. Secondarily, the length of the procedure and cosmetic results will be compared.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: When participating, patients will undergo 3 additional outpatient clinic visits. Study visits will be combined with regular visits where possible, including the first postoperative visit after 7-10 days and either the 6 week or 3 month visit.

ELIGIBILITY:
Inclusion Criteria:

* Female sex.
* 18 years or older.
* Indication for mastectomy.

Exclusion Criteria:

* Patients undergoing breast conserving therapy
* Patients undergoing direct breast reconstruction
* Patients undergoing modified radical mastectomy
* Unable to comprehend implications and extent of study and sign for informed consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 361 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Complications requiring an intervention | 3 months
  The main study parameter is the incidence of complications requiring interventions in both groups. This consists of:
  * Clinically significant seroma, requiring aspirations in the case of:
    * Pain or discomfort for the patient caused by large amounts of seroma characterised by tenderness of the skin.
    * Signs of infection (redness, swelling, pain).
    * Signs of delayed wound healing (wound breakdown, necrosis, seroma leakage).
  * Surgical site infections, requiring oral/iv antibiotics or surgical drainage.
  * Bleeding complications, requiring re-intervention, aspiration or surgical debridement.

SECONDARY OUTCOMES:
Surgery time | during surgery
  surgery time in minutes
Cosmetic outcome | 3 months
  • Cosmetic results measured using a numeric rating score (NRS) from 0-10, in which 0 equals very dissatisfied with the cosmetic results and 10 equals very satisfied with the results.

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland MC, Sittard, Limbrug, Netherlands

IPD SHARING:
Plan to Share IPD: No